CLINICAL TRIAL: NCT02607982
Title: Long-term Results of Definitive Concurrent Chemoradiotherapy Using Paclitaxel Plus Oxaliplatin in Unresectable Locally Advanced Esophageal Cancer.
Brief Title: CCRT for Esophageal Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Cancer Hospital (Other)
Responsible Party: Principal Investigator, Shixiu Wu, MD, Hangzhou Cancer Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangzhouCH03
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Esophageal Cancer; Concurrent Chemoradiotherapy; Oxaliplatin; Paclitaxel
Keywords: Esophageal cancer; Concurrent chemoradiotherapy; Oxaliplatin; Paclitaxel; Survival; Toxicity
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Concurrent Chemoradiotherapy Arm (Experimental): Radiotherapy was delivered with a daily fraction of 2.0 Gy to a total dose of 60 Gy over 6 weeks. Concurrent paclitaxel (135mg/m², d1) and oxaliplatin (125mg/ m², d1) were administered on Days 1 and Day 29 of radiotherapy.
  Interventions: Drug: Paclitaxel; Drug: Oxaliplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Paclitaxel — PTX 135 mg/m2 was administered intravenously over 3 hours on Day 1 and Day 29 with standard premedications.
Drug: Oxaliplatin — oxaliplatin (125mg/ m²) was given as a 2 hours infusion. Chemotherapy was started concurrently with radiation on day 1.
Radiation: Radiotherapy — Radiotherapy was given concurrently on the first day of the first cycle of chemotherapy. The GTV received 60Gy (30 fractions at 2Gy per fraction) and CTV was 40 Gy (20 fractions at 2Gy per fraction). Radiotherapy was delivered in three-dimensional conformal technique (3D-CRT) and no intensity-modulated radiotherapy was used.

SUMMARY:
This study aimed at assessing the efficiency and safety of concurrent chemoradiotherapy (CCRT) using paclitaxel (PTX) plus oxaliplatin (OHP) in unresectable locally advanced esophageal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically or histologically confirmed esophageal carcinoma
2. Age of 20 -80
3. ECOG performance status: 0-1;
4. No treatments prior to enrollment;
5. At least one measurable lesion on CT, MRI or esophageal barium exam;
6. Normal functions of heart, lung, liver, kidney and bone marrow
7. Blood exams qualified for chemotherapy, which included hemoglobulin ≥9 g/dl, neutrophil ≥1.5×109/L and platelet (PLT) ≥100×109/L, creatinine ≤1.5 UNL
8. Informed consent signed

Exclusion Criteria:

1. Prior treatments of chemotherapy or irradiation;
2. Poor bone marrow, liver and kidney functions, which would make chemotherapy intolerable;
3. Contraindication for irradiation: complete obstruction of esophagus, deep esophageal ulcer, fistula to mediastinum, or haematemesis;
4. Participating in other clinical trials;
5. Pregnancy, breast feeding, or not adopting birth control;
6. Clinically significant and uncontrolled major medical conditions including but not limited to: active uncontrolled infection, symptomatic congestive heart failure, Unstable angina pectoris or cardiac arrhythmia, psychiatric illness/ social situation that would limit compliance with study requirements; any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities
7. The subject has had another active malignancy within the past five years except for cervical cancer in site, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-01; Primary Completion 2014-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
response rate | week 4
  Response rate was done after 4 weeks following the last radiotherapy session.

SECONDARY OUTCOMES:
Survival outcome | year 0- year 5
  Progression-free survival (PFS) was calculated from the date of CCRT initiation to the date of documented failure (local recurrence or metastasis occurrence) or the date of the last follow-up for those remaining. Overall survival (OS) was determined as the time (in months) between the first day of therapy and the last follow-up or the date of death.
Toxicity | year 0- year 5
  Acute toxicities and late toxicities based on the common toxicity criteria for adverse events version 3.0 (CTCAEv3.0).

REFERENCES:
- [Background] Zhang P, Xie CY, Wu SX. [Concurrent chemoradiation with paclitaxel and platinum for locally advanced esophageal cancer]. Zhonghua Zhong Liu Za Zhi. 2007 Oct;29(10):773-7. Chinese. PMID 18396692